CLINICAL TRIAL: NCT00749879
Title: A Phase I, Open-Label, Randomized, Single-Center, Unblinded, Single-Dose, Five-Way Crossover Study of the Safety and PK Properties of Proellex®
Brief Title: Crossover Study of the Safety and PK Properties of Proellex®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ZP-008
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-01

CONDITIONS: Pharmacokinetics
Keywords: PK; Pharmacokinetics
MeSH Terms: interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 25 mg AMCC fed (Experimental): 25 mg Proellex capsule formulated with AMCC coarse microcrystalline cellulose
  Fed State
  Interventions: Drug: Proellex
- 25 mg AMCC fasting (Experimental): 25 mg Proellex capsule formulated with AMCC coarse microcrystalline cellulose
  Fasting State
  Interventions: Drug: Proellex
- 50 mg AMCC fed (Experimental): 2, 25 mg Proellex capsules formulated with AMCC coarse microcrystalline cellulose
  Fed State
  Interventions: Drug: Proellex
- 50 mg AMCC fasting (Experimental): 2, 25 mg Proellex capsules formulated with AMCC coarse microcrystalline cellulose
  Fasting State
  Interventions: Drug: Proellex
- 50 mg SMCC fasting (Experimental): 2, 25 mg Proellex capsules formulated with SMCC microcrystalline cellulose
  Fasting State
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Proellex — 25 mg capsule administered once orally after subjects have been fed; 25 mg capsule administered once orally while subjects are fasting; 2, 25 mg capsules administered once orally after subjects have been fed; 2, 25 mg capsules administered once orally while subjects are fasting; and 2, 25 mg capsules administered once orally while subjects are fasting
  Other Names: Telapristone acetate

SUMMARY:
Study to evaluate the PK of 25 mg and 50 mg of Proellex from 2 different suppliers in the fed and fasting states.

DETAILED DESCRIPTION:
This study is intended to evaluate the pharmacokinetic properties of two doses (25 mg and 50 mg) of Proellex® formulated with microcrystalline cellulose (MCC) from 2 different suppliers in the fed and fasting states.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to speak, read, and understand English and be willing and able to provide written informed consent in English on an Institutional Review Board (IRB)
* Premenopausal women aged 18-34, inclusive, with body mass index between 18 and 35, inclusive
* Women of child-bearing potential must be willing to use effective non-hormonal, double-barrier method contraception during the study period and for a minimum of 30 days after discontinuation of the study medication. Women who have had a hysterectomy will be allowed into the study
* Must have a negative urine pregnancy test at screening
* Able to swallow gelatin capsules
* Medically normal subjects with no significant abnormal findings at the screening physical examination as evaluated by the Principal Investigator that would interfere with the subject participating this study
* Must have agreed to not attempt to become pregnant at any time during study participation or for 30 days thereafter
* Other inclusion criteria may apply

Exclusion Criteria:

* Symptomatic uterine fibroids or endometriosis
* Past or present history of any significant cardiovascular, renal, or hepatic disease requiring ongoing medical therapy or clinical intervention
* Past or present history of thrombophlebitis, thromboembolic disorders, or cerebrovascular accident
* Abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Principal Investigator
* Significant organ abnormality or disease (based on the Principal Investigator's judgment) that would in the opinion of the Principal Investigator exclude the subject from participating
* Other exclusion criteria may apply

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-08-11 (Actual); Primary Completion 2008-10-23 (Actual); Study Completion 2008-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (1):
- Healthcare Discoveries Inc., San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 17 participants, 4 did not meet inclusion/exclusion criteria, and 1 participant enrolled as a spare was not needed, resulting in their involvement in the study being terminated. The remaining 12 participants completed all five study treatments of Proellex.
Pre-assignment Details: Each of the 12 participants were randomly assigned a unique sequence of the following 5 following open-label treatments of Proellex
  * 25 mg formulated with AMCC (fed state)
  * 25 mg formulated with AMCC (fasting state)
  * 50 mg formulated with AMCC (fed state)
  * 50 mg formulated with AMCC (fasting state)
  * 50 mg formulated with SMCC (fasting state)
Groups:
- Proellex: in randomly assigned sequences, all study participants received 5 open-label treatments of Proellex: 25 mg Proellex capsule formulated with AMCC coarse microcrystalline cellulose Fed State Proellex; 25 mg capsule administered once orally after subjects have been fed; 25 mg capsule administered once orally while subjects are fasting; 2, 25 mg capsules administered once orally after subjects have been fed; 2, 25 mg capsules administered once orally while subjects are fasting; and 2, 25 mg capsules administered once orally while subjects are fasting
Period: Overall Study
Arm/Group | Proellex
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled
Groups:
- All Subjects: All subjects enrolled
Arm/Group | All Subjects
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Proellex
Description: Maximum observed concentration of Proellex
Time Frame: Up to 72 hours post-dose
Population: 12 subjects received all 5 treatments
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 50 mg AMCC Fed: Two, 25 mg Proellex capsules formulated with AMCC coarse microcrystalline cellulose Fed State
- 50 mg AMCC Fasting: Two, 25 mg Proellex capsules formulated with AMCC coarse microcrystalline cellulose Fasting State
- 50 mg SMCC Fasting: Two, 25 mg Proellex capsules formulated with SMCC microcrystalline cellulose Fasting State
Arm/Group | 25 mg AMCC Fed | 25 mg AMCC Fasting | 50 mg AMCC Fed | 50 mg AMCC Fasting | 50 mg SMCC Fasting
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng/mL | 485.6 (151.3) | 876.7 (201.9) | 912.9 (157.6) | 1322.5 (154.5) | 1346.7 (148.5)

2. Primary Outcome: AUC0-last of Proellex
Description: Area under the plasma concentration curve from time 0 to the last measurable plasma concentration time point, up to 72 hours.
Time Frame: Up to 72 hours post dose
Population: All 12 subjects received each treatment
Measure: Mean (Standard Deviation); unit: ng/mL*hour
Arm/Group | 25 mg AMCC Fed | 25 mg AMCC Fasting | 50 mg AMCC Fed | 50 mg AMCC Fasting | 50 mg SMCC Fasting
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng/mL*hour | 6142.1 (2845.9) | 5765.7 (3036.6) | 11094.2 (4209.0) | 9252.0 (4217.5) | 9576.2 (4328.3)

3. Primary Outcome: Tmax of Proellex
Description: Time to maximum plasma occurrence of Cmax
Time Frame: Up to 72 hours post dose
Population: All 12 subjects received each treatment
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 25 mg AMCC Fed | 25 mg AMCC Fasting | 50 mg AMCC Fed | 50 mg AMCC Fasting | 50 mg SMCC Fasting
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Hours | 2.6 (0.6) | 0.8 (0.2) | 2.6 (1.0) | 0.9 (0.4) | 0.7 (0.2)

4. Primary Outcome: AUC0-infinity of Proellex
Description: Area under the plasma concentration curve from time 0 to extrapolated to infinity, calculated by summing the area under the curve from time zero to the time of the last quantifiable concentration
Time Frame: Up to 72 hours post dose
Population: All 12 subjects received each treatment
Measure: Mean (Standard Deviation); unit: ng/mL*hour
Arm/Group | 25 mg AMCC Fed | 25 mg AMCC Fasting | 50 mg AMCC Fed | 50 mg AMCC Fasting | 50 mg SMCC Fasting
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng/mL*hour | 7039.8 (3715.6) | 6897.0 (4440.7) | 13014.9 (6753.2) | 11271.6 (6726.6) | 11804.8 (7186.9)

5. Primary Outcome: Terminal Elimination Half-life (T1/2) of Proellex
Description: Time to maximum plasma occurrence of T1/2, calculated as ln(2)/Elimination rate constant.
Time Frame: Up to 72 hours post dose
Population: All 12 subjects received each treatment
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 25 mg AMCC Fed | 25 mg AMCC Fasting | 50 mg AMCC Fed | 50 mg AMCC Fasting | 50 mg SMCC Fasting
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Hours | 22.1 (8.2) | 25.2 (10.4) | 23.8 (10.8) | 26.7 (11.8) | 27.5 (11.9)

ADVERSE EVENTS:
Arm/Group | 25 mg AMCC Fed | 25 mg AMCC Fasting | 50 mg AMCC Fed | 50 mg AMCC Fasting | 50 mg SMCC Fasting
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12 | 4/12 | 7/12 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg AMCC Fed (N=12) | 25 mg AMCC Fasting (N=12) | 50 mg AMCC Fed (N=12) | 50 mg AMCC Fasting (N=12) | 50 mg SMCC Fasting (N=12)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pelvi pain NOS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oligomenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights